CLINICAL TRIAL: NCT03828617
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF 3 LOTS OF 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN PNEUMOCOCCAL VACCINE-NAÏVE ADULTS 18 THROUGH 49 YEARS OF AGE
Brief Title: Trial to Evaluate the Safety and Immunogenicity of 3 Lots of 20-valent Pneumococcal Conjugate Vaccine in Pneumococcal Vaccine-Naïve Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B7471008
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 20vPnC Lot 1 (Experimental): 20vPnC Lot 1
  Interventions: Biological: 20vPnC
- 20vPnC Lot 2 (Experimental): 20vPnC Lot 2
  Interventions: Biological: 20vPnC
- 20vPnC Lot 3 (Experimental): 20vPnC Lot 3
  Interventions: Biological: 20vPnC
- 13vPnC (Active Comparator): 13vPnC
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 20vPnC — 20vPnC
  Arms: 20vPnC Lot 1
Biological: 20vPnC — 20vPnC
  Arms: 20vPnC Lot 2
Biological: 20vPnC — 20vPnC
  Arms: 20vPnC Lot 3
Biological: 13vPnC — Pneumococcal conjugate vaccine
  Arms: 13vPnC

SUMMARY:
This is a Phase 3, randomized, double-blind study with a 4-arm parallel design. Adults 18 through 49 years of age with no history of pneumococcal vaccination will be randomized in a 2:2:2:1 ratio to receive a single dose of: 20vPnC Lot 1; 20vPnC Lot 2; 20vPnC Lot 3; or 13vPnC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥18 and <50 years of age.
2. Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including adults with preexisting stable disease, defined as disease not requiring significant change in therapy in the previous 6 weeks or hospitalization for worsening disease within 12 weeks before receipt of investigational product.
3. Female subject of childbearing potential or male subject who is able to father children, and willing to use a highly effective method of contraception as outlined in this protocol for at least 28 days after the dose of investigational product; or female subject not of childbearing potential or male subject not able to father children.

Exclusion Criteria:

1. Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.
2. Serious chronic disorder including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the subject from participating in the study.
3. History of microbiologically proven invasive disease caused by S pneumoniae.
4. Pregnant female subjects or breastfeeding female subjects (known or suspected).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1710 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (21):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Kaiser Permanente South Sacramento, Sacramento, California
  - Kaiser Permanente San Jose, San Jose, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Accel Research Sites - Clinical Research Unit, DeLand, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East West Medical Research Institute, Honolulu, Hawaii
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Rochester Clinical Research, Inc., Rochester, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Omega Medical Research, Warwick, Rhode Island
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - Benchmark Research, Austin, Texas
  - J. Lewis Research, Inc. /Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. /Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sabharwal C, Sundaraiyer V, Peng Y, Moyer L, Belanger TJ, Gessner BD, Jodar L, Jansen KU, Gruber WC, Scott DA, Watson W. Immunogenicity of a 20-valent pneumococcal conjugate vaccine in adults 18 to 64 years old with medical conditions and other factors that increase risk of pneumococcal disease. Hum Vaccin Immunother. 2022 Nov 30;18(6):2126253. doi: 10.1080/21645515.2022.2126253. Epub 2022 Nov 11. PMID 36368038
- [Derived] Klein NP, Peyrani P, Yacisin K, Caldwell N, Xu X, Scully IL, Scott DA, Jansen KU, Gruber WC, Watson W. A phase 3, randomized, double-blind study to evaluate the immunogenicity and safety of 3 lots of 20-valent pneumococcal conjugate vaccine in pneumococcal vaccine-naive adults 18 through 49 years of age. Vaccine. 2021 Sep 7;39(38):5428-5435. doi: 10.1016/j.vaccine.2021.07.004. Epub 2021 Jul 24. PMID 34315611
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1718 participants were enrolled, out of which only 1710 were randomized. There were 8 participants who were enrolled (signed informed consent document) but were not randomized into the study as the randomization system had reached the pre-specified capacity.
Groups:
- 20vPnC Lot 1: Participants were randomized to receive a single 0.5 milliliter (mL) intramuscular injection of 20-valent pneumococcal vaccine (20vPnC) from Lot 1 on Day 1. Participants were followed up to 6 months after vaccination.
- 20vPnC Lot 2: Participants were randomized to receive a single 0.5 mL intramuscular injection of 20vPnC from Lot 2 on Day 1. Participants were followed up to 6 months after vaccination.
- 20vPnC Lot 3: Participants were randomized to receive a single 0.5 mL intramuscular injection of 20vPnC from Lot 3 on Day 1. Participants were followed up to 6 months after vaccination.
- 13vPnC: Participants were randomized to receive a single 0.5 mL intramuscular injection of 13-valent pneumococcal vaccine (13vPnC) on Day 1. Participants were followed up to 6 months after vaccination.
Period: Overall Study
Arm/Group | 20vPnC Lot 1 | 20vPnC Lot 2 | 20vPnC Lot 3 | 13vPnC
Started | 489 | 490 | 486 | 245
Vaccinated | 488 | 489 | 486 | 245
Safety Population | 488 | 489 | 486 | 245
Evaluable Immunogenicity Population(EIP) | 463 | 473 | 456 | 232
Completed | 465 | 475 | 460 | 235
Not Completed | 24 | 15 | 26 | 10
Not completed — Lost to Follow-up | 22 | 12 | 23 | 7
Not completed — No longer met eligibility criteria | 0 | 1 | 1 | 3
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received 1 dose of any 20vPnC lot or 13vPnC and had safety follow-up after the vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20vPnC Lot 1 | 20vPnC Lot 2 | 20vPnC Lot 3 | 13vPnC | Total
Number analyzed (Participants) | 488 | 489 | 486 | 245 | 1708
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (9.17) | 35.7 (9.03) | 34.9 (9.05) | 35.0 (8.70) | 35.3 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331 | 316 | 324 | 144 | 1115
  Male | 157 | 173 | 162 | 101 | 593
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 58 | 56 | 29 | 191
  Not Hispanic or Latino | 434 | 427 | 427 | 215 | 1503
  Unknown or Not Reported | 6 | 4 | 3 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 9 | 5 | 4 | 23
  Asian | 13 | 17 | 17 | 12 | 59
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 2 | 6
  Black or African American | 87 | 88 | 97 | 44 | 316
  White | 367 | 351 | 350 | 173 | 1241
  More than one race | 6 | 13 | 13 | 5 | 37
  Unknown or Not Reported | 8 | 10 | 3 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 10 Days After Vaccination
Description: Local reactions were recorded using an electronic diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm) and severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity). Data for this outcome measure was planned to be analyzed for the pooled 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) and 13vPnC group.
Time Frame: Within 10 days after vaccination
Population: Safety population included all participants who received 1 dose of any 20vPnC lot or 13vPnC and had safety follow-up after the vaccination. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled 20vPnC: Participants were randomized to receive a single 0.5 mL intramuscular injection of 20vPnC from any of the lots 1, 2 or 3 on Day 1. Participants were followed up to 6 months after vaccination.
Arm/Group | Pooled 20vPnC | 13vPnC
Number analyzed (Participants) | 1456 | 243
percentage of participants
  Redness: Any | 7.0 [5.7 to 8.4] | 6.2 [3.5 to 10.0]
  Redness: Mild | 3.9 [3.0 to 5.0] | 3.3 [1.4 to 6.4]
  Redness: Moderate | 2.6 [1.9 to 3.6] | 2.9 [1.2 to 5.8]
  Redness: Severe | 0.5 [0.2 to 1.0] | 0 [0.0 to 1.5]
  Swelling: Any | 8.5 [7.1 to 10.1] | 8.6 [5.4 to 12.9]
  Swelling: Mild | 5.4 [4.3 to 6.7] | 5.3 [2.9 to 9.0]
  Swelling: Moderate | 2.9 [2.1 to 3.9] | 3.3 [1.4 to 6.4]
  Swelling: Severe | 0.2 [0.0 to 0.6] | 0 [0.0 to 1.5]
  Pain at the injection site: Any | 78.7 [76.5 to 80.8] | 75.7 [69.8 to 81.0]
  Pain at the injection site: Mild | 50.0 [47.4 to 52.6] | 46.5 [40.1 to 53.0]
  Pain at the injection site: Moderate | 27.5 [25.3 to 29.9] | 27.6 [22.1 to 33.6]
  Pain at the injection site: Severe | 1.2 [0.7 to 1.9] | 1.6 [0.5 to 4.2]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events fever, fatigue, headache, muscle pain, joint pain were recorded by using an electronic diary. Fever was defined as greater than or equal to (>=) 38.0 degree Celsius (C) and categorized to >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Fatigue, headache, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity). Data for this outcome measure was planned to be analyzed for the pooled 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) and 13vPnC group.
Time Frame: Within 7 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled 20vPnC | 13vPnC
Number analyzed (Participants) | 1456 | 243
percentage of participants
  Fever: >=38.0 degree C (Any) | 1.2 [0.7 to 1.9] | 0.8 [0.1 to 2.9]
  Fever: >=38.0 degree C to 38.4 degree C | 0.8 [0.4 to 1.3] | 0.4 [0.0 to 2.3]
  Fever: >38.4 degree C to 38.9 degree C | 0.3 [0.1 to 0.7] | 0.4 [0.0 to 2.3]
  Fever: >38.9 degree C to 40.0 degree C | 0.2 [0.0 to 0.6] | 0 [0.0 to 1.5]
  Fever: >40.0 degree C | 0 [0.0 to 0.3] | 0 [0.0 to 1.5]
  Fatigue: Any | 47.6 [45.0 to 50.2] | 43.6 [37.3 to 50.1]
  Fatigue: Mild | 24.7 [22.5 to 27.0] | 24.3 [19.0 to 30.2]
  Fatigue: Moderate | 21.2 [19.1 to 23.4] | 17.7 [13.1 to 23.1]
  Fatigue: Severe | 1.7 [1.1 to 2.5] | 1.6 [0.5 to 4.2]
  Headache: Any | 36.2 [33.7 to 38.7] | 37.9 [31.7 to 44.3]
  Headache: Mild | 22.6 [20.5 to 24.8] | 27.2 [21.7 to 33.2]
  Headache: Moderate | 12.0 [10.4 to 13.8] | 9.9 [6.4 to 14.3]
  Headache: Severe | 1.6 [1.0 to 2.4] | 0.8 [0.1 to 2.9]
  Muscle pain: Any | 62.1 [59.5 to 64.6] | 60.5 [54.0 to 66.7]
  Muscle pain: Mild | 38.5 [36.0 to 41.0] | 38.7 [32.5 to 45.1]
  Muscle pain: Moderate | 22.5 [20.4 to 24.8] | 19.8 [14.9 to 25.3]
  Muscle pain: Severe | 1.1 [0.6 to 1.8] | 2.1 [0.7 to 4.7]
  Joint pain: Any | 16.8 [14.9 to 18.8] | 14.0 [9.9 to 19.0]
  Joint pain: Mild | 10.0 [8.5 to 11.6] | 7.8 [4.8 to 11.9]
  Joint pain: Moderate | 6.5 [5.2 to 7.8] | 5.3 [2.9 to 9.0]
  Joint pain: Severe | 0.4 [0.2 to 0.9] | 0.8 [0.1 to 2.9]

3. Primary Outcome: Percentage of Participants With Any Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in study participants who received study vaccine without regard to possibility of causal relationship. Data for this outcome measure was planned to be analyzed for the pooled 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) and 13vPnC group.
Time Frame: Within 1 month after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled 20vPnC | 13vPnC
Number analyzed (Participants) | 1463 | 245
percentage of participants | 6.8 [5.6 to 8.3] | 5.3 [2.9 to 8.9]

4. Primary Outcome: Percentage of Participants With Any Serious Adverse Events (SAEs) Within 6 Months After Vaccination
Description: An SAE was any untoward medical occurrence at any dose that results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect or that is considered to be an important medical event. Data for this outcome measure was planned to be analyzed for the pooled 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) and 13vPnC group.
Time Frame: Within 6 month after vaccination
Population: Safety population includes all participants who received 1 dose of any 20vPnC lot or 13vPnC and had safety follow-up after the vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled 20vPnC | 13vPnC
Number analyzed (Participants) | 1463 | 245
percentage of participants | 0.7 [0.3 to 1.3] | 0 [0.0 to 1.5]

5. Primary Outcome: Percentage of Participants With Any Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 6 Months After Vaccination
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects. Data for this outcome measure was planned to be analyzed for the pooled 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) and 13vPnC group.
Time Frame: Within 6 months after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pooled 20vPnC | 13vPnC
Number analyzed (Participants) | 1463 | 245
percentage of participants | 1.0 [0.6 to 1.7] | 2.0 [0.7 to 4.7]

6. Primary Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at 1 Month After Vaccination
Description: OPA titers were determined for serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F. OPA titer was expressed as reciprocal of the highest serum dilution. OPA GMTs and 2-sided 95% CIs were calculated. Data for this outcome measure were planned to be analyzed for the 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) only.
Time Frame: 1 month after vaccination
Population: EIP: participants who received randomized vaccine, had blood collection within 27 to 49 days after vaccination (Visit 2), had at least 1 valid and determinate OPA titer for any serotype at Visit 2, and had no other major protocol deviations. Here, "Number analyzed" = participants evaluable for this outcome measure at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 20vPnC Lot 1 | 20vPnC Lot 2 | 20vPnC Lot 3
Number analyzed (Participants) | 463 | 473 | 456
titer
  Serotype 1: number analyzed (Participants) | 462 | 470 | 454
  Serotype 1 | 199.5 [173.5 to 229.6] | 175.1 [152.5 to 201.0] | 164.6 [143.1 to 189.3]
  Serotype 3: number analyzed (Participants) | 458 | 469 | 451
  Serotype 3 | 47.3 [42.7 to 52.4] | 46.8 [42.3 to 51.8] | 43.1 [38.9 to 47.8]
  Serotype 4: number analyzed (Participants) | 455 | 468 | 451
  Serotype 4 | 1499.7 [1288.3 to 1745.6] | 1568.2 [1350.2 to 1821.4] | 1505.6 [1294.4 to 1751.3]
  Serotype 5: number analyzed (Participants) | 457 | 466 | 450
  Serotype 5 | 125.8 [108.6 to 145.7] | 135.6 [117.3 to 156.7] | 116.8 [100.9 to 135.2]
  Serotype 6A: number analyzed (Participants) | 454 | 468 | 446
  Serotype 6A | 4654.1 [4033.0 to 5371.0] | 3748.3 [3255.7 to 4315.4] | 3330.4 [2885.1 to 3844.6]
  Serotype 6B: number analyzed (Participants) | 458 | 469 | 453
  Serotype 6B | 4403.3 [3832.6 to 5059.0] | 4349.9 [3796.4 to 4984.1] | 3907.3 [3401.4 to 4488.3]
  Serotype 7F: number analyzed (Participants) | 452 | 464 | 441
  Serotype 7F | 1820.6 [1588.5 to 2086.5] | 1865.6 [1629.7 to 2135.7] | 1875.7 [1632.6 to 2154.9]
  Serotype 9V: number analyzed (Participants) | 454 | 467 | 446
  Serotype 9V | 5120.4 [4464.6 to 5872.7] | 4604.1 [4024.4 to 5267.5] | 4921.7 [4292.4 to 5643.2]
  Serotype 14: number analyzed (Participants) | 455 | 467 | 450
  Serotype 14 | 2240.2 [1965.4 to 2553.5] | 2091.2 [1839.9 to 2376.8] | 2001.9 [1760.4 to 2276.5]
  Serotype 18C: number analyzed (Participants) | 455 | 465 | 449
  Serotype 18C | 3903.7 [3339.6 to 4563.2] | 4450.7 [3818.1 to 5188.0] | 4221.7 [3615.8 to 4929.2]
  Serotype 19A: number analyzed (Participants) | 451 | 465 | 450
  Serotype 19A | 1457.8 [1287.5 to 1650.6] | 1528.1 [1353.2 to 1725.6] | 1434.4 [1267.8 to 1623.0]
  Serotype 19F: number analyzed (Participants) | 455 | 466 | 452
  Serotype 19F | 524.5 [450.7 to 610.3] | 529.2 [455.6 to 614.6] | 549.0 [472.2 to 638.3]
  Serotype 23F: number analyzed (Participants) | 459 | 471 | 454
  Serotype 23F | 1416.1 [1182.4 to 1696.1] | 1547.5 [1294.9 to 1849.2] | 1434.6 [1197.8 to 1718.1]
  Serotype 8: number analyzed (Participants) | 435 | 448 | 436
  Serotype 8 | 1595.0 [1402.7 to 1813.7] | 1345.9 [1185.9 to 1527.6] | 1624.3 [1430.4 to 1844.5]
  Serotype 10A: number analyzed (Participants) | 399 | 418 | 410
  Serotype 10A | 6328.1 [5407.7 to 7405.2] | 5692.6 [4890.2 to 6626.6] | 5962.2 [5121.3 to 6941.1]
  Serotype 11A: number analyzed (Participants) | 394 | 399 | 399
  Serotype 11A | 8656.2 [7308.4 to 10252.5] | 6728.5 [5693.2 to 7952.0] | 8720.3 [7408.6 to 10264.1]
  Serotype 12F: number analyzed (Participants) | 418 | 418 | 411
  Serotype 12F | 8563.0 [7321.5 to 10015.0] | 7907.5 [6764.8 to 9243.3] | 7412.4 [6331.8 to 8677.4]
  Serotype 15B: number analyzed (Participants) | 392 | 426 | 402
  Serotype 15B | 7342.8 [6108.1 to 8827.2] | 6356.9 [5325.0 to 7588.7] | 7018.9 [5853.8 to 8416.1]
  Serotype 22F: number analyzed (Participants) | 367 | 392 | 384
  Serotype 22F | 12507.5 [10318.3 to 15161.1] | 11213.4 [9337.1 to 13466.9] | 12728.6 [10571.7 to 15325.5]
  Serotype 33F: number analyzed (Participants) | 391 | 401 | 409
  Serotype 33F | 10745.7 [9042.0 to 12770.5] | 10328.2 [8737.0 to 12209.3] | 10418.2 [8815.3 to 12312.5]
Statistical Analysis 1: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 1: Geometric mean ratios (GMRs) (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% confidence intervals (CIs); Test type: Equivalence — Lots were considered equivalent if each of the pairwise 2-sided 95% CIs for the GMRs of OPA titers was contained in the interval (0.5, 2.0); Geometric Mean Ratio (GMR) = 1.14, 95% CI 2-sided [0.95 to 1.37]
Statistical Analysis 2: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 3: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio (GMR) = 1.01, 95% CI 2-sided [0.88 to 1.16]
Statistical Analysis 3: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 4: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.96, 95% CI 2-sided [0.78 to 1.17]
Statistical Analysis 4: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 5: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.77 to 1.12]
Statistical Analysis 5: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 6A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.24, 95% CI 2-sided [1.03 to 1.50]
Statistical Analysis 6: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 6B: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.85 to 1.21]
Statistical Analysis 7: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 7F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.98, 95% CI 2-sided [0.82 to 1.17]
Statistical Analysis 8: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 9V: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.11, 95% CI 2-sided [0.93 to 1.33]
Statistical Analysis 9: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 14: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.07, 95% CI 2-sided [0.90 to 1.27]
Statistical Analysis 10: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 18C: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.88, 95% CI 2-sided [0.72 to 1.07]
Statistical Analysis 11: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 19A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.95, 95% CI 2-sided [0.81 to 1.12]
Statistical Analysis 12: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 19F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.81 to 1.21]
Statistical Analysis 13: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 23F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.92, 95% CI 2-sided [0.72 to 1.16]
Statistical Analysis 14: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 8: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.19, 95% CI 2-sided [1.00 to 1.40]
Statistical Analysis 15: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 10A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.11, 95% CI 2-sided [0.91 to 1.36]
Statistical Analysis 16: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 11A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.29, 95% CI 2-sided [1.03 to 1.60]
Statistical Analysis 17: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 12F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.08, 95% CI 2-sided [0.88 to 1.33]
Statistical Analysis 18: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 15B: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.16, 95% CI 2-sided [0.91 to 1.46]
Statistical Analysis 19: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 22F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.12, 95% CI 2-sided [0.87 to 1.43]
Statistical Analysis 20: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 2; Serotype 33F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 2) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.04, 95% CI 2-sided [0.83 to 1.30]
Statistical Analysis 21: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 1: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.21, 95% CI 2-sided [1.01 to 1.46]
Statistical Analysis 22: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 3: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.10, 95% CI 2-sided [0.96 to 1.26]
Statistical Analysis 23: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 4: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.00, 95% CI 2-sided [0.82 to 1.22]
Statistical Analysis 24: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 5: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.08, 95% CI 2-sided [0.89 to 1.31]
Statistical Analysis 25: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 6A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.40, 95% CI 2-sided [1.16 to 1.69]
Statistical Analysis 26: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 6B: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.13, 95% CI 2-sided [0.94 to 1.35]
Statistical Analysis 27: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 7F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.97, 95% CI 2-sided [0.81 to 1.16]
Statistical Analysis 28: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 9V: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.04, 95% CI 2-sided [0.87 to 1.25]
Statistical Analysis 29: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 14: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.12, 95% CI 2-sided [0.94 to 1.33]
Statistical Analysis 30: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 18C: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.92, 95% CI 2-sided [0.75 to 1.13]
Statistical Analysis 31: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 19A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.02, 95% CI 2-sided [0.86 to 1.20]
Statistical Analysis 32: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 19F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.96, 95% CI 2-sided [0.78 to 1.17]
Statistical Analysis 33: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 23F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.78 to 1.25]
Statistical Analysis 34: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 8: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.98, 95% CI 2-sided [0.83 to 1.16]
Statistical Analysis 35: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 10A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.06, 95% CI 2-sided [0.87 to 1.30]
Statistical Analysis 36: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 11A: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.80 to 1.24]
Statistical Analysis 37: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 12F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.16, 95% CI 2-sided [0.94 to 1.42]
Statistical Analysis 38: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 15B: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.82 to 1.33]
Statistical Analysis 39: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 22F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.98, 95% CI 2-sided [0.77 to 1.26]
Statistical Analysis 40: Comparison: 20vPnC Lot 1 vs 20vPnC Lot 3; Serotype 33F: GMRs (ratio of GMTs for 20vPnC Lot 1 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.03, 95% CI 2-sided [0.82 to 1.29]
Statistical Analysis 41: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 1: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.06, 95% CI 2-sided [0.89 to 1.28]
Statistical Analysis 42: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 3: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.09, 95% CI 2-sided [0.95 to 1.24]
Statistical Analysis 43: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 4: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.04, 95% CI 2-sided [0.85 to 1.27]
Statistical Analysis 44: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 5: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.16, 95% CI 2-sided [0.96 to 1.41]
Statistical Analysis 45: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 6A: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.13, 95% CI 2-sided [0.93 to 1.36]
Statistical Analysis 46: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 6B: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.11, 95% CI 2-sided [0.93 to 1.33]
Statistical Analysis 47: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 7F: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.83 to 1.19]
Statistical Analysis 48: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 9V: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.94, 95% CI 2-sided [0.78 to 1.12]
Statistical Analysis 49: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 14: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.04, 95% CI 2-sided [0.88 to 1.24]
Statistical Analysis 50: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 18C: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.86 to 1.29]
Statistical Analysis 51: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 19A: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.07, 95% CI 2-sided [0.91 to 1.25]
Statistical Analysis 52: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 19F: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.96, 95% CI 2-sided [0.79 to 1.17]
Statistical Analysis 53: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 23F: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.08, 95% CI 2-sided [0.85 to 1.37]
Statistical Analysis 54: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 8: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.83, 95% CI 2-sided [0.70 to 0.98]
Statistical Analysis 55: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 10A: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.95, 95% CI 2-sided [0.78 to 1.17]
Statistical Analysis 56: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 11A: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.62 to 0.96]
Statistical Analysis 57: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 12F: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 1.07, 95% CI 2-sided [0.87 to 1.31]
Statistical Analysis 58: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 15B: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.91, 95% CI 2-sided [0.71 to 1.15]
Statistical Analysis 59: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 22F: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.88, 95% CI 2-sided [0.69 to 1.12]
Statistical Analysis 60: Comparison: 20vPnC Lot 2 vs 20vPnC Lot 3; Serotype 33F: GMRs (ratio of GMTs for 20vPnC Lot 2 to Lot 3) and 2-sided 95% CIs; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.79 to 1.24]

7. Secondary Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From Before Vaccination to 1 Month After Vaccination
Description: Fold rises are the ratios of the 1 month after vaccination to before vaccination OPA titers. OPA GMFRs from before to 1 month after vaccination were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F. Data for this outcome measure was planned to be analyzed for the 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) only.
Time Frame: Before vaccination to 1 month after vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 20vPnC Lot 1 | 20vPnC Lot 2 | 20vPnC Lot 3
Number analyzed (Participants) | 463 | 473 | 456
fold rise
  Serotype 1: number analyzed (Participants) | 460 | 468 | 454
  Serotype 1 | 20.2 [17.6 to 23.1] | 17.8 [15.6 to 20.3] | 17.3 [15.0 to 19.8]
  Serotype 3: number analyzed (Participants) | 456 | 462 | 449
  Serotype 3 | 5.0 [4.4 to 5.5] | 5.0 [4.5 to 5.5] | 4.6 [4.1 to 5.1]
  Serotype 4: number analyzed (Participants) | 441 | 450 | 435
  Serotype 4 | 77.6 [63.8 to 94.4] | 94.7 [79.4 to 112.9] | 81.0 [67.0 to 97.8]
  Serotype 5: number analyzed (Participants) | 455 | 463 | 450
  Serotype 5 | 8.7 [7.5 to 10.0] | 9.4 [8.2 to 10.7] | 8.0 [6.9 to 9.1]
  Serotype 6A: number analyzed (Participants) | 436 | 451 | 429
  Serotype 6A | 157.2 [132.6 to 186.3] | 119.6 [100.5 to 142.3] | 128.4 [107.6 to 153.1]
  Serotype 6B: number analyzed (Participants) | 423 | 442 | 424
  Serotype 6B | 72.5 [59.9 to 87.8] | 75.4 [62.9 to 90.4] | 70.5 [58.1 to 85.6]
  Serotype 7F: number analyzed (Participants) | 422 | 424 | 401
  Serotype 7F | 18.3 [15.5 to 21.7] | 19.5 [16.5 to 23.0] | 19.0 [16.1 to 22.5]
  Serotype 9V: number analyzed (Participants) | 398 | 409 | 387
  Serotype 9V | 25.4 [21.1 to 30.7] | 23.3 [19.4 to 27.9] | 21.6 [17.7 to 26.4]
  Serotype 14: number analyzed (Participants) | 426 | 436 | 434
  Serotype 14 | 18.2 [14.8 to 22.3] | 16.3 [13.2 to 20.0] | 18.1 [14.6 to 22.3]
  Serotype 18C: number analyzed (Participants) | 435 | 448 | 439
  Serotype 18C | 80.4 [63.9 to 101.2] | 95.0 [76.6 to 117.7] | 79.9 [63.8 to 100.0]
  Serotype 19A: number analyzed (Participants) | 443 | 456 | 440
  Serotype 19A | 35.9 [29.9 to 43.2] | 39.1 [32.4 to 47.1] | 41.8 [34.9 to 50.2]
  Serotype 19F: number analyzed (Participants) | 450 | 458 | 448
  Serotype 19F | 14.0 [12.0 to 16.5] | 14.7 [12.6 to 17.2] | 15.4 [13.1 to 18.0]
  Serotype 23F: number analyzed (Participants) | 452 | 458 | 445
  Serotype 23F | 99.5 [80.4 to 123.1] | 125.1 [102.4 to 152.7] | 120.9 [97.9 to 149.5]
  Serotype 8: number analyzed (Participants) | 416 | 429 | 418
  Serotype 8 | 38.3 [31.3 to 46.8] | 38.8 [32.1 to 46.9] | 46.1 [37.9 to 56.0]
  Serotype 10A: number analyzed (Participants) | 350 | 368 | 370
  Serotype 10A | 20.8 [16.6 to 26.1] | 19.0 [15.2 to 23.7] | 20.2 [15.9 to 25.6]
  Serotype 11A: number analyzed (Participants) | 319 | 321 | 332
  Serotype 11A | 6.9 [5.4 to 8.9] | 5.0 [3.9 to 6.4] | 5.3 [4.2 to 6.7]
  Serotype 12F: number analyzed (Participants) | 390 | 389 | 376
  Serotype 12F | 175.5 [141.3 to 217.9] | 174.6 [140.8 to 216.7] | 175.7 [141.6 to 218.1]
  Serotype 15B: number analyzed (Participants) | 364 | 395 | 369
  Serotype 15B | 112.5 [83.8 to 150.9] | 84.2 [64.5 to 110.0] | 91.7 [69.4 to 121.3]
  Serotype 22F: number analyzed (Participants) | 322 | 357 | 338
  Serotype 22F | 83.8 [59.2 to 118.6] | 63.3 [46.8 to 85.7] | 77.8 [56.8 to 106.6]
  Serotype 33F: number analyzed (Participants) | 338 | 357 | 362
  Serotype 33F | 8.3 [6.7 to 10.4] | 8.6 [7.0 to 10.6] | 7.4 [6.0 to 9.1]

8. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 4 -Fold Rise in Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Titers From Before Vaccination to 1 Month After Vaccination
Description: Percentage of participants with a >=4-fold rise in serotype-specific pneumococcal OPA titers from before vaccination to 1 month after vaccination along with corresponding 2-sided 95% CIs were calculated for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F. Data for this outcome measure was planned to be analyzed for the 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) only.
Time Frame: Before vaccination to 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Lot 1 | 20vPnC Lot 2 | 20vPnC Lot 3
Number analyzed (Participants) | 463 | 473 | 456
percentage of participants
  Serotype 1: number analyzed (Participants) | 460 | 468 | 454
  Serotype 1 | 83.7 [80.0 to 87.0] | 82.9 [79.2 to 86.2] | 82.4 [78.6 to 85.8]
  Serotype 3: number analyzed (Participants) | 456 | 462 | 449
  Serotype 3 | 56.1 [51.4 to 60.8] | 57.8 [53.1 to 62.3] | 53.0 [48.3 to 57.7]
  Serotype 4: number analyzed (Participants) | 441 | 450 | 435
  Serotype 4 | 85.0 [81.4 to 88.2] | 87.6 [84.1 to 90.5] | 86.2 [82.6 to 89.3]
  Serotype 5: number analyzed (Participants) | 455 | 463 | 450
  Serotype 5 | 65.7 [61.2 to 70.1] | 67.2 [62.7 to 71.4] | 65.3 [60.7 to 69.7]
  Serotype 6A: number analyzed (Participants) | 436 | 451 | 429
  Serotype 6A | 94.5 [91.9 to 96.4] | 93.1 [90.4 to 95.3] | 93.0 [90.2 to 95.2]
  Serotype 6B: number analyzed (Participants) | 423 | 442 | 424
  Serotype 6B | 90.3 [87.1 to 93.0] | 91.4 [88.4 to 93.8] | 89.2 [85.8 to 91.9]
  Serotype 7F: number analyzed (Participants) | 422 | 424 | 401
  Serotype 7F | 76.8 [72.4 to 80.7] | 76.7 [72.3 to 80.6] | 80.0 [75.8 to 83.9]
  Serotype 9V: number analyzed (Participants) | 398 | 409 | 387
  Serotype 9V | 79.1 [74.8 to 83.0] | 79.5 [75.2 to 83.3] | 75.7 [71.1 to 79.9]
  Serotype 14: number analyzed (Participants) | 426 | 436 | 434
  Serotype 14 | 70.0 [65.4 to 74.3] | 67.7 [63.0 to 72.0] | 67.7 [63.1 to 72.1]
  Serotype 18C: number analyzed (Participants) | 435 | 448 | 439
  Serotype 18C | 83.0 [79.1 to 86.4] | 88.2 [84.8 to 91.0] | 84.5 [80.8 to 87.8]
  Serotype 19A: number analyzed (Participants) | 443 | 456 | 440
  Serotype 19A | 81.7 [77.8 to 85.2] | 81.8 [77.9 to 85.2] | 85.5 [81.8 to 88.6]
  Serotype 19F: number analyzed (Participants) | 450 | 458 | 448
  Serotype 19F | 74.0 [69.7 to 78.0] | 76.2 [72.0 to 80.0] | 75.2 [71.0 to 79.2]
  Serotype 23F: number analyzed (Participants) | 452 | 458 | 445
  Serotype 23F | 85.6 [82.0 to 88.7] | 88.2 [84.9 to 91.0] | 88.8 [85.5 to 91.5]
  Serotype 8: number analyzed (Participants) | 416 | 429 | 418
  Serotype 8 | 82.0 [77.9 to 85.5] | 82.3 [78.3 to 85.8] | 82.5 [78.5 to 86.1]
  Serotype 10A: number analyzed (Participants) | 350 | 368 | 370
  Serotype 10A | 74.9 [70.0 to 79.3] | 74.5 [69.7 to 78.8] | 70.8 [65.9 to 75.4]
  Serotype 11A: number analyzed (Participants) | 319 | 321 | 332
  Serotype 11A | 52.4 [46.7 to 57.9] | 48.0 [42.4 to 53.6] | 42.2 [36.8 to 47.7]
  Serotype 12F: number analyzed (Participants) | 390 | 389 | 376
  Serotype 12F | 91.8 [88.6 to 94.3] | 93.1 [90.1 to 95.4] | 91.5 [88.2 to 94.1]
  Serotype 15B: number analyzed (Participants) | 364 | 395 | 369
  Serotype 15B | 81.6 [77.2 to 85.4] | 82.0 [77.9 to 85.7] | 81.0 [76.7 to 84.9]
  Serotype 22F: number analyzed (Participants) | 322 | 357 | 338
  Serotype 22F | 79.8 [75.0 to 84.1] | 82.1 [77.7 to 85.9] | 81.4 [76.8 to 85.4]
  Serotype 33F: number analyzed (Participants) | 338 | 357 | 362
  Serotype 33F | 62.7 [57.3 to 67.9] | 62.7 [57.5 to 67.8] | 62.7 [57.5 to 67.7]

9. Secondary Outcome: Percentage of Participants With Serotype-specific Opsonophagocytic Activity (OPA) Titers Greater Than or Equal to Lower Limit of Quantitation (>= LLOQ) at 1 Month After Vaccination
Description: The percentage of participants with OPA titers >=LLOQ were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. Data for this outcome measure was planned to be analyzed for the 20vPnC vaccine groups (20vPnC Lots 1, 2 and 3) only.
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Lot 1 | 20vPnC Lot 2 | 20vPnC Lot 3
Number analyzed (Participants) | 463 | 473 | 456
percentage of participants
  Serotype 1: number analyzed (Participants) | 462 | 470 | 454
  Serotype 1 | 91.8 [88.9 to 94.1] | 92.8 [90.0 to 94.9] | 91.0 [87.9 to 93.4]
  Serotype 3: number analyzed (Participants) | 458 | 469 | 451
  Serotype 3 | 89.7 [86.6 to 92.4] | 89.6 [86.4 to 92.2] | 88.9 [85.6 to 91.7]
  Serotype 4: number analyzed (Participants) | 455 | 468 | 451
  Serotype 4 | 97.6 [95.7 to 98.8] | 97.0 [95.0 to 98.4] | 97.1 [95.1 to 98.5]
  Serotype 5: number analyzed (Participants) | 457 | 466 | 450
  Serotype 5 | 80.3 [76.4 to 83.9] | 84.3 [80.7 to 87.5] | 81.3 [77.4 to 84.8]
  Serotype 6A: number analyzed (Participants) | 454 | 468 | 446
  Serotype 6A | 99.1 [97.8 to 99.8] | 98.1 [96.4 to 99.1] | 98.2 [96.5 to 99.2]
  Serotype 6B: number analyzed (Participants) | 458 | 469 | 453
  Serotype 6B | 97.6 [95.7 to 98.8] | 99.6 [98.5 to 99.9] | 98.9 [97.4 to 99.6]
  Serotype 7F: number analyzed (Participants) | 452 | 464 | 441
  Serotype 7F | 94.7 [92.2 to 96.6] | 94.0 [91.4 to 96.0] | 96.6 [94.5 to 98.1]
  Serotype 9V: number analyzed (Participants) | 454 | 467 | 446
  Serotype 9V | 98.5 [96.8 to 99.4] | 98.9 [97.5 to 99.7] | 98.2 [96.5 to 99.2]
  Serotype 14: number analyzed (Participants) | 455 | 467 | 450
  Serotype 14 | 98.9 [97.5 to 99.6] | 99.4 [98.1 to 99.9] | 97.8 [96.0 to 98.9]
  Serotype 18C: number analyzed (Participants) | 455 | 465 | 449
  Serotype 18C | 96.9 [94.9 to 98.3] | 98.1 [96.4 to 99.1] | 98.7 [97.1 to 99.5]
  Serotype 19A: number analyzed (Participants) | 451 | 465 | 450
  Serotype 19A | 99.3 [98.1 to 99.9] | 100.0 [99.2 to 100.0] | 99.3 [98.1 to 99.9]
  Serotype 19F: number analyzed (Participants) | 455 | 466 | 452
  Serotype 19F | 91.2 [88.2 to 93.6] | 91.0 [88.0 to 93.4] | 90.7 [87.6 to 93.2]
  Serotype 23F: number analyzed (Participants) | 459 | 471 | 454
  Serotype 23F | 94.3 [91.8 to 96.3] | 95.8 [93.5 to 97.4] | 94.9 [92.5 to 96.8]
  Serotype 8: number analyzed (Participants) | 435 | 448 | 436
  Serotype 8 | 98.6 [97.0 to 99.5] | 99.1 [97.7 to 99.8] | 99.1 [97.7 to 99.7]
  Serotype 10A: number analyzed (Participants) | 399 | 418 | 410
  Serotype 10A | 99.7 [98.6 to 100.0] | 99.0 [97.6 to 99.7] | 99.3 [97.9 to 99.8]
  Serotype 11A: number analyzed (Participants) | 394 | 399 | 399
  Serotype 11A | 99.2 [97.8 to 99.8] | 99.5 [98.2 to 99.9] | 99.5 [98.2 to 99.9]
  Serotype 12F: number analyzed (Participants) | 418 | 418 | 411
  Serotype 12F | 99.0 [97.6 to 99.7] | 99.3 [97.9 to 99.9] | 99.0 [97.5 to 99.7]
  Serotype 15B: number analyzed (Participants) | 392 | 426 | 402
  Serotype 15B | 99.0 [97.4 to 99.7] | 98.6 [97.0 to 99.5] | 99.3 [97.8 to 99.8]
  Serotype 22F: number analyzed (Participants) | 367 | 392 | 384
  Serotype 22F | 99.7 [98.5 to 100.0] | 99.2 [97.8 to 99.8] | 99.5 [98.1 to 99.9]
  Serotype 33F: number analyzed (Participants) | 391 | 401 | 409
  Serotype 33F | 99.0 [97.4 to 99.7] | 98.8 [97.1 to 99.6] | 98.5 [96.8 to 99.5]

ADVERSE EVENTS:
Time Frame: Local reactions: within 10 days after vaccination (systematic assessment), Systemic events: within 7 days after vaccination (systematic assessment), Non serious AEs: up to 1 month after vaccination, SAEs: up to 6 months after vaccination
Description: Event may be categorized as serious in 1 participant and non-SAE in another participant or 1 participant may have experienced both SAE and non-SAE. Safety population was used. Because the primary safety objective was to describe the safety profile of 20vPnC and not the safety profile for each lot of 20vPnC,the safety data for 20vPnC in this study are reported as pooled data. The pooled data represent the safety population of 20vPnC in this study and are summarized with the 13vPnC control group.
Arm/Group | Pooled 20vPnC | 13vPnC
All-Cause Mortality (participants affected / at risk) | 0/1463 | 0/245
Serious Adverse Events (participants affected / at risk) | 10/1463 | 0/245
Other Adverse Events (participants affected / at risk) | 1275/1463 | 206/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled 20vPnC (N=1463) | 13vPnC (N=245)
Splenic cyst (Blood and lymphatic system disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled 20vPnC (N=1463) | 13vPnC (N=245)
Fatigue (General disorders) | 693 | 106
Injection site erythema (REDNESS) (General disorders) | 102 | 15
Injection site pain (PAIN) (General disorders) | 1146 | 184
Injection site swelling (SWELLING) (General disorders) | 124 | 21
Pyrexia (FEVER) (General disorders) | 18 | 2
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 245 | 34
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 904 | 147
Headache (Nervous system disorders) | 527 | 92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT03828617/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03828617/SAP_003.pdf